CLINICAL TRIAL: NCT05119491
Title: Relation Between Pulmonary Function Tests and Ultrasonographic Changes of Asymptomatic Anterior Chest Wall Joints in Rheumatoid Arthritis Patients
Brief Title: Relation Between Pulmonary Function Tests and Ultrasonographic Chest Joints
Acronym: Ultrasound
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Waleed Mansour, Ass prof, Zagazig University
Other Study IDs: 7039
Record Dates: First submitted 2021-10-07; First posted 2021-11-15 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Restrictive Lung Disease
MeSH Terms: interventions — Spirometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases ultra sound and spirometry: observation by ultra sound and spirometry for cases
  Interventions: Device: uitrasonography and spirometry
- heathy subjects ultra sound and spirometry: observation ultra sound and spirometry for control heathy subjects
  Interventions: Device: uitrasonography and spirometry

INTERVENTIONS:
Device: uitrasonography and spirometry — chest uitrasonography and spirometry

SUMMARY:
Ultrasonography can detect different changes in anterior chest wall (ACW) joints in patients with Rheumatoid arthritis (RA) even before being clinically manifested. Airways ,pleura, lung parenchyma and vascular compartment all may be attacked by RA. This study was aiming at detecting the relation between ultrasonographic changes of asymptomatic ACW joints and pulmonary function tests (PFTs) in patients with RA.

DETAILED DESCRIPTION:
1. Clinical assessment:

   Patients and controls were examined in supine position with elbows placed in contact with the body. The anterior chest wall joints (CWJ) which include the right and left sternoclavicular (SCJ) and manubriosternal (MSJ) joints were evaluated for presence/absence of spontaneous pain, pain evoked by digital pressure, swelling, and redness of skin.

   Rheumatoid disease activity was assessed clinically using: disease activity score (DAS28 ESR)] and Functional status assessment by health assessment questionnaire (HAQ) .

   Chest expansion was measured with a tape measure placed circumferentially around the chest wall at the fourth intercostal space.
2. US assessment:

   Ultrasonographic B examination (mode and Doppler power mode) of the 3 joints were performed by an experienced rheumatologist. All patients were examined using B-mode (gray scale) real-time MSUS (F37; Hitachi-Aloka, Japan) interfaced with a 10-18-MHz linear array transducer. For each patient and control subject, US examination included a longitudinal section of the left and right SCJ and the MSJ, followed by a cross-section in case erosion was detected. During the examination, synovitis (hypo echoic intracapsular incompressible area with or without Doppler flow), joint effusion (compressible anechoic intracapsular area, absence of Doppler flow), erosion (disruption of the cortical bone line displayed in 2 perpendicular axes), joint space narrowing (reduction of the joint space), ankylosis (complete loss of joint space), or Doppler signal (power Doppler signal) were investigated.

   PD parameters were as follow: Pulse repetition frequency (PRF) was adjusted at the lowest permissible value to maximize sensitivity. This setting resulted in PRF from 500 Hz to 750 Hz. Flow was additionally demonstrated in 2 planes and confirmed by pulsed wave Doppler spectrum to exclude artifacts.

   Computed Tomography (HRCT) was done on the chest to exclude any interstitial lung disease that may affect chest expansion and restrictive PFTs.
3. Pulmonary function tests:

PFTs was done with a Sensormedics Vmax229 system (Sensormedics, Yorba Linda, California, USA) and included measurement of the forced expiratory volume in1 second (FEV1), forced vital capacity (FVC), and the ratio of forced expiratory volume in 1 second to the forced vital capacity(FEV1/FVC).

The study was approved by the Institutional Review Board at the Faculty of Medicine, Zagazig University Hospitals. It has been carried out in accordance with the code of ethics of the world medical association (Declaration of Helsinki 1964) for studies involving humans. A written informed consent was obtained from each participant.

Methods:

Aim: To detect the relation between ultrasonographic changes of asymptomatic ACW joints and pulmonary function tests (PFTs) in patients with RA.

Study design and setting: An observational case control study.

ELIGIBILITY:
Inclusion Criteria:

* rheumatoid arthritis patients

Exclusion Criteria:

* other respiratory diseases

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: rheumatoid arthritis patients
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-03-21 (Actual)

PRIMARY OUTCOMES:
This study is a trial to find correlation between US detected abnormalities in anterior chest wall joints and (FEV1,FVC,FEV1/FVC ) in Rh A patients | about 2 years
  observation

CONTACTS AND LOCATIONS:
Locations (1):
- zagazigU, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
research